CLINICAL TRIAL: NCT07041541
Title: Clinical Evaluation of Gingivalstat Approach Compared to Conventional Esthetic Crown Lengthening on the Stability of The Gingival Margin in Patients With Altered Passive Eruption. A Randomized Clinical Trial.
Brief Title: Clinical Evaluation of Gingivalstat Approach Compared to Conventional Esthetic Crown Lengthening on the Stability of The Gingival Margin in Patients With Altered Passive Eruption.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Elganayni, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Composite stops after ECL
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Gummy Smile; Altered Passive Eruption of Teeth; Healthy Participants
Keywords: Gummy Smile; Altered Passive Eurption; Esthetic Crown Lengthening; GingivalStat Approach

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Gingival Stat approach -- Composite stops after ECL surgery) (Experimental): Steps 1-6 as Active Comparator group + 7. Resin composite wil be placed on the cervical third of the teeth, following the CEJ anatomy, to act as a gingival stabilizer to guide the early remodelling of tissues.
  8. Removal of sutures and composite after two weeks.
  Interventions: Procedure: Esthetic Crown Lengthening using GingivalStat approach
- Control group (Conventional ECL surgery) (Active Comparator): 1. Following the administration of local anaesthesia, a submarginal internal bevelled incision using 15c blade will be carried out, from canine to canine. The distance from the gingival margin will be based on how much soft tissue needs to be removed to meet the ideal tooth proportion.
  2. Intrasulcular incision will be done in the buccal aspect and papilla region for removal of tissue collar.
  3. A full thickness mucoperiosteal flap will be elevated using mucoperiosteal elevator, without bypassing the MGJ.
  4. To obtain a 3 mm distance between CEJ and bone, osteoctomy wil be carried out from line angle to line angle using high speed hand piece with end-cutting bur.
  5. Osteoplasty using round bur, maybe done to reduce bone thickness and obtain adequate anatomical profile.
  6. After the flap is repositioned, interrupted sutures using Polypropylene 5-0 will be used to adapt and suture the flap in its new position.
  Interventions: Procedure: Esthetic Crown Lengthening

INTERVENTIONS:
Procedure: Esthetic Crown Lengthening — Conventional Esthetic Crown Lengthening
  Arms: Control group (Conventional ECL surgery)
Procedure: Esthetic Crown Lengthening using GingivalStat approach — Esthetic Crown Lengthening using GingivalStat approach (composite stops)
  Arms: Interventional group (Gingival Stat approach -- Composite stops after ECL surgery)

SUMMARY:
When performing crown lengthening surgery, especially in the esthetic zone, the positional stability of gingival tissues is considered a prime important goal. The rebound of gingival margins after surgery can result in compromising the esthetic outcome and patient satisfaction. It was proven throughout the literature that there are many factors that may influence the stability of gingival margin position after surgery such as: the surgical technique being performed, experience of the clinician, periodontal phenotype and distance of flap with respect to the alveolar crest.

DETAILED DESCRIPTION:
A "gummy smile" or excessive gingival display (EGD) is when at least 3-5 mm of gingiva is visible. It is viewed as unnatural or unsightly, and in order to have the best outcome, cosmetic periodontal recontouring is frequently necessary. It is considered the treatment of choice for excessive gingival display, or "Gummy smile,". Many causes of gummy smiles have been found, including altered passive eruption, short upper lip, dentoalveolar extrusion, abnormal vertical bone growth, and a combination of some of these.

Altered passive eruption is when the gingival margin is located incisal to the cervical convexity of the crown and away from the cemento-enamel junction of the tooth. It is considered the most frequent related factor, accounting for between 12.1 and 35.8% of excessive gingival display cases that have been identified, according to evidence.

Considering esthetic crown lengthening (ECL) surgery, the goal is to restore the gingival harmony and symmetry by reestablishing the proper clinical crown length. However, stability of the periodontal tissues after ECL is a crucial aspect that can be jeopardized the treatment outcome of the treated region. In particular, gingival margin rebound can impair aesthetics and have an impact on the health of periodontal tissue

Predicting the amount of tissue rebound after esthetic crown lengthening surgery is still controversial. According to literature, there is a tendency to have a gingival regrowth from the immediate postoperative level for up to 3 months. It has been also confirmed that rebound of gingival margin most likely occurs during the first three months following surgery. Another study found that the gingival margin had coronal migration may continue for up to 6-12 months after surgery.

Based on current evidence, gingival margin rebound is a major issue that happens after performing crown lengthening surgery. To avoid this, GingivalStat approach has been proposed to guide the tissue after surgery to remodel early at a predetermined position and avoid the re-growth of gingiva in a coronal direction. It appears to be producing earlier stability. The current study aims to investigate the influence of GingivalStat following crown lengthening versus conventional crown lengthening, in terms of stability of gingival margin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Altered Passive Eruption Subtype B presenting altered alveolar bone crest-CEJ relationship according to Coslet's et al. classification.
2. Patients free of systemic diseases.
3. Patients aged between 18 to 60 years old.
4. Patients maintaining good oral hygiene with full-mouth plaque and bleeding scores <15%.
5. Patients should be committed to the post-operative care regime, including oral hygiene practices, and follow-up visits.

Exclusion Criteria:

1. Areas in which the remaining amount of keratinized gingiva after the submarginal incision will be less than 3 mm.
2. Patients with periodontal disease.
3. Smokers.
4. Pregnant women.
5. Patients on medication that may interfere with healing (corticosteroids, bisphosphonate, Chemo/radiotherapy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the gingival margin | Baseline, immediate post operative, 2 weeks, 3 months and 6 months
  Gingival margin position wil be measured using UNC periodontal probe + stent. Grooves will be made in the stent to standardize probe direction and localization. Each tooth will be assessed on the mesio-buccal, mid-buccal, and disto-buccal aspect at baseline, immediate post operative, 2 weeks, 3 months, and 6 months.
Stability of relative gingival margin position | Baseline, immediate postoperative, 2 weeks, 3 months and 6 months
  Gingival margin position will be measured using Intra-oral digital Scan (IOS). It will be measured at baseline, immediately after surgery, 2 weeks, 3 months and 6 months. Scans will be superimposed to detect all changes throughout the follow up period.

SECONDARY OUTCOMES:
Pink Esthetic Score by blinded assessment | At 3 months and 6 months
  It is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable is assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Postsurgical pain assessment | At two weeks.
  Readings will be recorded by the patient for the first 14 days after the surgery using the VAS which is a descriptive numerical rating scale of 0 to 10.
  0 = No pain 1-3= Mild pain 4-6 = Moderate pain (bearable) 7-10 = Severe pain (unbearable)
Patient satisfaction | Two weeks, three months and six months
  A 3-item questionnaire will be given to the patients to be answered using a 7-point answer scale for assessing their satisfaction with the whole procedure and the results of the procedure performed.
Cost effectiveness | At six months.
  It will be calculated using an equation to correlate the procedural time, cost of the materials used against the clinical outcomes.
Procedural Time | At the surgery
  It will be recorded in minutes using a stopwatch to measure the difference in the procedural time between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt